CLINICAL TRIAL: NCT04766346
Title: Nutritional Supplementation in Children Aged 1-3 Years Experiencing Growth Concerns: a Prospective, Single-arm, Open-label, Interventional Study
Brief Title: Nutritional Supplementation in Children Aged 1-3 Years Experiencing Growth Concerns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20.09.INF
Record Dates: First submitted 2020-12-16; First posted 2021-02-23 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Growth; Learning; Toddlers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional Supplement (Experimental): The NS is a fortified cow's milk-based product provided in powdered form.
  Interventions: Other: Fortified Cow's Milk-Based Oral Nutritional Supplement

INTERVENTIONS:
Other: Fortified Cow's Milk-Based Oral Nutritional Supplement — The NS is a fortified cow's milk-based product provided in powdered form that provides the appropriate amount of energy and protein to promote growth in children.

SUMMARY:
This open-label clinical trial will gain evidence of the effect of an oral Nutritional Supplement (NS) to help improve catch-up growth and support learning skills in children with growth concerns.

ELIGIBILITY:
INCLUSION CRITERIA

1. Evidence of a personally signed and dated informed consent document indicating that the child's parent(s) / legally acceptable representative (LAR) has been informed of all pertinent aspects of the study.
2. Child was full-term at birth (i.e., ≥ 37 completed weeks of gestation with a birth weight of ≥ 2.5 kg and ≤ 4.5 kg).
3. Child is age 12 - 36 months and generally healthy (acute illness in a minor condition which are common in childhood such as viral or bacterial infection e.g. conjunctivitis, otitis media, upper/lower respiratory tract infection, gastroenteritis, hand foot & mouth disease at time of enrolment is permitted).
4. Children whose parents show some concern about their child's growth, such as child is too thin for his or her length/height, child has experienced recent rapid weight loss or failure to gain weight or length/height, or child's growth curve shows a downward trajectory of growth velocity
5. Child has a weight-for-length/height ≤ 25th percentile as per WHO growth charts.
6. Parents agree to feed their child a nutritional supplement in addition to normal diet.
7. Child's parent(s) / guardian can be contacted directly by telephone or email throughout the study.
8. Child's parent is of legal age of consent, must understand the informed consent form and other study documents, and is willing and able to fulfill the requirements of the study protocol.

EXCLUSION CRITERIA

1. Child is currently breastfed or is consuming breast milk
2. Child has known or suspected cows' milk protein intolerance / allergy, lactose intolerance, soy intolerance / allergy, fish oil intolerance / allergy, or other food allergies that impact diet.
3. Child fed vegan, vegetarian, or vegetarian plus fish diets in which milk products are excluded
4. Child has chronic illness or other disease including any condition that impacts feeding or growth
5. Child having any congenital malformation (e.g., gastrointestinal tract atresia) or surgery sequelae (e.g., short bowel syndrome) potentially affecting feeding or growth
6. Child has been diagnosed with Infantile anorexia nervosa
7. Child has other medical or psychiatric condition that, in the judgement of the investigator, would make the child inappropriate for entry into the study.
8. Child or child's parent(s) not willing and/or not able to comply with scheduled visits and the requirements of the study protocol.
9. Child of any investigational site staff member or Nestlé employee directly involved in the conduct of the trial.
10. Child is currently participating in or has participated in another clinical trial within 4 weeks prior to enrolment.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
The primary objective of this clinical trial is to to assess the effect of NS on weight gain and linear growth. | Day 1 to Day 113
  The primary endpoint is the change in weight-for-length/height z-score

SECONDARY OUTCOMES:
Weight | Day 1, Day 22, Day 43, Day 64, Day 85, Day 113
  Measurement of Weight in grams
Length/height | Day 1, Day 22, Day 43, Day 64, Day 85, Day 113
  Measurement of length/height in cms
Triceps skin fold thickness | Day 1, Day 22, Day 43, Day 64, Day 85, Day 113
  Measurement of triceps skinfold thickness
Sub-scapular skinfold thickness | Day 1, Day 22, Day 43, Day 64, Day 85, Day 113
  Measurement of sub-scapular skinfold thickness in mm
Suprailiac skinfold thickness | Day 1, Day 22, Day 43, Day 64, Day 85, Day 113
  Measurement of suprailiac skinfold thickness in mm
BMI | Day 1, Day 22, Day 43, Day 64, Day 85, Day 113
  BMI will be calculated and expressed in Kg/m2
Z scores and percentiles | Day 1, Day 22, Day 43, Day 64, Day 85, Day 113
  1) Sex-age-specific weight, length/height, BMI and triceps and subscapular skinfold thickness percentiles and Z-scores calculated according to WHO standards. 2) Changes from baseline in sex-age-specific percentiles and Z-scores
Nutrient intake | Day 22, Day 43, Day 113
  Nutrient intake from 3-day Food Intake Diaries that will be completed at home for two weekdays and 1 weekend day
Learning skills | Day 1, Day 113
  Learning Scores derived from the Ages and Stages Questionnaire, Third Edition (ASQ-3) (with a focus on communication and problem-solving skills)
Temperament and behavior | Day 1, Day 113
  Temperament and behaviour scores from the Early Childhood Behavior Questionnaire- Short Form (ECBQ-SF) completed. The ECBQ-SF has 107 questions and assesses dimensions of temperament such as activity Level/Energy, attentional Focusing, attentional Shifting, cuddliness, discomfort, fear, frustration, high-intensity Pleasure, impulsivity, inhibitory Control, low-intensity Pleasure, motor Activation, perceptual Sensitivity, positive Anticipation, sadness, shyness, sociability and soothability.The scale items ask parents to report on the frequency of specific behaviours in frequently occurring contexts on a 7 point likert scale ranging from never to always.
Child and parent well-being reported from the parents' perspective | Day 1, Day 113
  Child health-related quality of life scores assessed using the Infant and Toddler Quality of Life Questionnaire Short Form (ITQOL-SF47). The ITQOL-SF47 has 47 questions and assesses domains such as the overall health, physical abilities, growth and development, bodily pain/discomfort, temperament and moods, general health perceptions, parent impact - emotional, parent impact - time and family cohesion with a score of 0 (worst) to 100 (best) for each of these domains.
Product acceptance | Day 22, Day 64, Day 113
  Product acceptance scores from the Toddler Milk Satisfaction Questionnaire
Product acceptance including child-liking and post-ingestive effects | Day 22, Day 64, Day 113
  Primary facial expression valence and child heart rate variability derived from the ANURA for Research (smartphone app) while child is consuming one serving of the NS

OTHER OUTCOMES:
Safety assessment | Day -7 to Day 113 + 30
  Data from standard AE reporting (including common illnesses) for safety assessment from date of ICF signing through 30 days after the last day of NS intake.
Sick days | Day -7 to Day 113 + 30
  Total number of sick days
Concomittant medications and treatment | Day -7 to Day 113 + 30
  All concomitant medications / treatments used to treat illnesses and other conditions will be recorded (both dose and duration) through 30 days after the last day of NS intake.

CONTACTS AND LOCATIONS:
Locations (1):
- Las Piñas Doctors Hospital, Las Piñas, Philippines

IPD SHARING:
Plan to Share IPD: Undecided